CLINICAL TRIAL: NCT06788834
Title: Multimodal Prehabilitation in Cancer Surgery PROPOSE Trial (PRehabilitation in Oncological Patients undergOing SurgEry): A Randomized Trial
Brief Title: Multimodal Prehabilitation in Cancer Surgery
Acronym: PROPOSE-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Prof. Pasquale Sansone (Unknown); Prof. Eugenio Garofalo (Unknown); Prof. Tiziana Bove (Unknown); Dr. Claudia Brusasco (Unknown); Prof. Gabriele Baldini (Unknown); Dr. Nicola Passuello (Unknown); Dr. Monica Gualtierotti (Unknown); Prof. Luca Carlo Nespoli (Unknown)
Responsible Party: Principal Investigator, Marina Pieri, Doctor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PNRR-MCNT2-2023-12378183
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer Surgery
Keywords: Prehabilitation; Functional recovery; Relaxation; Exercise; Diet; Nutrition; Functional walking; Hospital stay; Multimodal prehabilitation program; Standard treatment; Anesthesiology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation (Experimental): The prehabilitation arm group will receive preoperative intervention which includes exercise training, nutritional therapy and anxiety reducing techniques, aimed at preventing or attenuating surgery-driven functional decline. This will be on top of Standard care treatment with application of ERAS pathways (Enhanced Recovery After Surgery).
  Interventions: Behavioral: Multimodal prehabilitation Program
- Control group (No Intervention): Standard care treatment with application of ERAS pathways (Enhanced Recovery After Surgery)

INTERVENTIONS:
Behavioral: Multimodal prehabilitation Program — A tailored intervention will be prescribed if specific physical, nutritional or psychological impairments will be identified during the assessment phase.
  Based on the data obtained during the multimodal assessment, different domains and levels of care will be prescribed, focusing on exercise training, and/or nutrition optimization, and/or distress-coping techniques. Different combinations of three domains will be utilized to maximize their synergistic anabolic effects. The duration of the program will be set at a minimum of three weeks.
  Arms: Prehabilitation

SUMMARY:
The PROPOSE RCT is a two-arm randomized controlled trial that will be conducted to test the efficacy of a personalized, multidisciplinary pre-operative prehabilitation program (preventive prehabilitation) to reduce serious complications and facilitate recovery after surgery in high-risk patients.

The multimodal prehabilitation program is a preoperative intervention that includes exercise training, nutritional therapy and anxiety reduction techniques, with the aim of preventing or mitigating the functional decline brought about by surgery. 400 patients scheduled for elective major abdominal (including urological), thoracic (including breast) or gynecological cancer surgery will be enrolled. They will be randomized (1:1 ratio) and assigned either to the intervention group (Prehabilitation) or to the control group, which will only be treated according to the usual standard of care within the Enhanced Recovery After Surgery (ERAS) pathways.

DETAILED DESCRIPTION:
The standard treatment for most solid cancer includes surgery and concurrent medical therapies, both of which have been shown to significantly improve prognosis. However, cancer treatments impose impactful physiological stress and have detrimental effects on acute and long-term health outcomes.

Physical, nutritional, and mental status can influence surgical outcomes, functional recovery and quality of life throughout the course of the disease.

The importance of postoperative rehabilitation on physical performance and recovery is well-recognized. However, the preoperative period provides a unique opportunity to address comorbidities and modifiable risk factors. In addition, the metabolic stress induced by neoadjuvant therapy has been documented to frequently result in muscle atrophy and diminished functional capacity. The recognition that selected risk factors of poor postoperative outcome can be modified has prompted clinicians to identify proactive interventions to facilitate the recovery process. In this context, prehabilitation, aimed at enhancing the patients' functional capacity to enable them to withstand the physiological stress of surgery, has emerged as a promising approach. Although the term prehabilitation is not novel, the concept of optimizing patients before acute stressor or treatment has gained attention over the last decade. Nonetheless, quantifiable evidence of its effectiveness has yet to be fully demonstrated.

This study is a multicenter randomized controlled trial to assess the efficacy of personalized procedure-specific prehabilitation programs on patient-centered surgical outcomes. A total of 400 patients will be recruited by systematic screening of patients scheduled for elective surgical procedures. All patients undergoing elective major abdominal (including urological), thoracic (including breast) or gynecological cancer surgery undergoing major cancer surgery will be screened for eligibility and those who meet the inclusion/exclusion criteria will be approached for consent. Research personnel will use a web-based randomization system to assign patients (1:1 ratio) to either the prehabilitation or control arm. Study personnel will also collect data on recruitment rates, with reasons for non-enrolment.

Eligible patients will be randomly assigned to 1 of 2 treatments:

1. multimodal prehabilitation program for at least three weeks started as soon as possible before surgery;
2. standard care.

The multimodal prehabilitation program will be individualized by carefully integrating and adapting various components to meet individual needs. The program will last at least three weeks (plus maintenance in case of delayed surgery), and will incorporate exercise training, nutritional therapy, and anxiety reduction techniques. After enrollment, patients will receive initial contact from trained personnel through telemedicine. To ensure personalized care, a comprehensive assessment will be conducted to identify specific physical, nutritional, or psychological challenges. Based on this assessment, a customized intervention plan will be prescribed to achieve tailored exercise training, optimized nutrition, and effective distress-coping strategies. All patients will be reassessed the day before surgery and 30 days after surgery. Based on the data obtained during the multimodal assessment, different domains and levels of care will be prescribed, focusing on exercise training, nutrition optimization, or distress-coping techniques-or a combination of these

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years);
* Scheduled for elective major abdominal (including urological), thoracic (including breast) or gynecological cancer surgery;
* Signed informed consent.

Exclusion Criteria:

A) Co-morbid medical, physical, and mental conditions interfering with the ability to complete study procedures, such as:

* Acute or unstable cardio-respiratory conditions (e.g., unstable angina or symptomatic severe aortic stenosis);
* Severe/end-stage organ diseases (e.g., cardiac failure NYHA functional classes III-IV, COPD FEV1 <50% pred, end-stage kidney or liver disease);
* American Society of Anesthesiologists (ASA) physical status classes 4-5;
* Disabling orthopedic and neuromuscular disease;
* Psychosis, dementia;
* Symptomatic anemia with a hemoglobin value < 7 gr/dl.

B) Patients with both optimal functional capacity (a Duke activity status index [DASI] score > 45) and optimal nutritional status (NRS-nutrition screening tool-score < 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of prehabilitation on severe postoperative complications among high-risk patients undergoing oncological surgery | 30 days after surgery
  The proportion of patients experiencing severe postoperative complications within 30 days after surgery defined as grade 3a or greater according to the Clavien-Dindo classification

SECONDARY OUTCOMES:
Time to Functional Recovery (TFR) | 30 days after surgery
  Faster return to basal functional preoperative capacity in treatment group
Lenght of hospital stay (LOS) | 30 days after surgery
  Reduction of lenght of hospital stay in treatment group
Days at home up to 30 days after surgery (DAH-30) | 30 days after surgery
  The mean number of days at home in the first 30 days after surgery will be compared between groups
Complication severity | 30 days after surgery
  Assess complication severity as measured by the Comprehensive Complication Index (CCI)
Proportion of patients returning to preoperative functional walking capacity | 30 days after surgery
  Improvement in the return to basal functional preoperative capacity
Self-reported activity status and generic health related quality of life | 30 days after surgery
  Assess quality of life in the first 30 days at home after surgery using the EuroQol-5 Dimension (EQ-5D-5L) questionnaire, a validated tool for evaluating health-related quality of life. The outcome will be reported as the mean EQ-5D-5L index score and the mean EQ-VAS score measured at 30 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Pieri, Medical Doctor, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (9):
- Italy (9):
  - Policlinico Universitario AOU Renato Dulbecco di Catanzaro, Catanzaro, Italy
  - AOU Careggi, Florence, Italy
  - Ospedale Galliera di Genova, Genova, Italy
  - ASSTN GOM Niguarda, Milan, Italy
  - IRCCS Ospedale San Gerardo dei Tintori, Monza, Italy
  - Ospedale Vanvitelli di Napoli, Napoli, Italy
  - AOPD Padova, Padua, Italy
  - Azienda sanitaria universitaria Friuli Centrale (ASU FC), Udine, Italy
  - IRCCS Ospedale San Raffaele, Milan, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colado JC, Pedrosa FM, Juesas A, Gargallo P, Carrasco JJ, Flandez J, Chupel MU, Teixeira AM, Naclerio F. Concurrent validation of the OMNI-Resistance Exercise Scale of perceived exertion with elastic bands in the elderly. Exp Gerontol. 2018 Mar;103:11-16. doi: 10.1016/j.exger.2017.12.009. Epub 2017 Dec 17. PMID 29262307
- [Background] Levett DZH, Jack S, Swart M, Carlisle J, Wilson J, Snowden C, Riley M, Danjoux G, Ward SA, Older P, Grocott MPW; Perioperative Exercise Testing and Training Society (POETTS). Perioperative cardiopulmonary exercise testing (CPET): consensus clinical guidelines on indications, organization, conduct, and physiological interpretation. Br J Anaesth. 2018 Mar;120(3):484-500. doi: 10.1016/j.bja.2017.10.020. Epub 2017 Nov 24. PMID 29452805
- [Background] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Background] Silver JK, Baima J. Cancer prehabilitation: an opportunity to decrease treatment-related morbidity, increase cancer treatment options, and improve physical and psychological health outcomes. Am J Phys Med Rehabil. 2013 Aug;92(8):715-27. doi: 10.1097/PHM.0b013e31829b4afe. PMID 23756434
- [Background] Lemanne D, Cassileth B, Gubili J. The role of physical activity in cancer prevention, treatment, recovery, and survivorship. Oncology (Williston Park). 2013 Jun;27(6):580-5. PMID 23909073
- [Background] Carli F. Physiologic considerations of Enhanced Recovery After Surgery (ERAS) programs: implications of the stress response. Can J Anaesth. 2015 Feb;62(2):110-9. doi: 10.1007/s12630-014-0264-0. Epub 2014 Dec 12. PMID 25501695